CLINICAL TRIAL: NCT02856360
Title: Changes in Footwear Comfort and Performance in High School Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Collaborators: Adidas International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-004
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Foot; Footwear
Keywords: Football; Cleats; Stiffness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Stiffness (Experimental): Shoe condition that has moderate stiffness
  Interventions: Other: Moderate Stiffness Footwear
- High Stiffness (Active Comparator): Shoe condition that has high stiffness
  Interventions: Other: High Stiffness Footwear

INTERVENTIONS:
Other: Moderate Stiffness Footwear — Standard moderately stiff footwear for typical high school football players will be randomly allocated to each group
  Arms: Moderate Stiffness
Other: High Stiffness Footwear — Standard highly stiff footwear for typical high school football players will be randomly allocated to each group
  Arms: High Stiffness

SUMMARY:
The objective of this proposal is to determine the effects of footwear stiffness on a large cohort of high school football players during a football season. The investigators expect that functional athlete groups will be developed, based on subject specific assessments (biomechanical, morphological, performance, comfort), and lead to important translational findings that may impact footwear modification and recommendation to a population of American football players. Two standard cleats will be randomized and provided during a season of high school football. Ratings of comfort, performance, and injury will be collected throughout the season.

ELIGIBILITY:
Inclusion Criteria:

* Participate on a club or school sponsored football team

Exclusion Criteria:

* Current injury that limits sport participation

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07; Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Footwear comfort rating using a 100mm visual analog scale | 3 months
  Validated subjective rating of footwear comfort scale. This will be collected weekly during the football season with the average rating utilized at the end of the season. The unit of measure is a 100mm visual analog scale.

SECONDARY OUTCOMES:
Injury incidence | 3 months
  Athletic trainer collected athletic exposures and lower extremity injuries will be collected weekly and combined to determine overall injury rates. The unit of measure is number of injuries per 1000 athletic exposures.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Biomechanics and Physiology Laboratory, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No